CLINICAL TRIAL: NCT00037323
Title: Framingham Offspring Study: Psychosocial Risk Factors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1162; R03HL067426 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression; Atrial Fibrillation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression; Atrial Fibrillation

SUMMARY:
To examine the relationship between psychosocial characteristics, health behaviors, and the development of coronary heart disease among participants in the Framingham Offspring Study.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Unique data sets of social, psychological, and behavioral measures were collected at the third examination of the Offspring Study from 1984 through 1987 (which results in 14 to 17 years of follow-up). Hypotheses for this research are focused toward understanding the sex and age differences in the effects these variables have on health endpoints. The research questions involve the prediction of three separate endpoints: incidence of coronary heart disease; the incidence and prognosis of atrial fibrillation; and total mortality. The analyses of psychosocial predictors for these outcomes are divided into four conceptual areas: 1) occupational status and strain, income, and employment status; 2) type A behavior, expressions of anger, hostility, and rate; 3) symptoms of depression, tension, anxiety, and feelings of aloneness; and 4) marital relationships and marital strain. These psychosocial variables will be analyzed jointly with the physiological risk factors collected at the same time to assess independence and interaction of effects. To date these psychosocial data have not been analyzed or published.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Study Completion 2003-10 (Actual)

REFERENCES:
- [Background] Eaker ED, Sullivan LM, Kelly-Hayes M, D'Agostino RB Sr, Benjamin EJ. Does job strain increase the risk for coronary heart disease or death in men and women? The Framingham Offspring Study. Am J Epidemiol. 2004 May 15;159(10):950-8. doi: 10.1093/aje/kwh127. PMID 15128607
- [Background] Eaker ED, Sullivan LM, Kelly-Hayes M, D'Agostino RB Sr, Benjamin EJ. Anger and hostility predict the development of atrial fibrillation in men in the Framingham Offspring Study. Circulation. 2004 Mar 16;109(10):1267-71. doi: 10.1161/01.CIR.0000118535.15205.8F. Epub 2004 Mar 1. PMID 14993133